CLINICAL TRIAL: NCT06675305
Title: Acute Effects of Beetroot Juice Ingestion on Cognitive Function and Neuromuscular Performance in Elite Female Taekwondo Athletes
Acronym: BEET_TAEKWONDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Collaborators: Universidad Complutense de Madrid (Other); University of Seville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ethics Committee: 22/172-E_TFM
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Dietary Supplements: Beetroot Juice Acute Supplementation; Dietary Supplement: Placebo Acute Supplementation
Keywords: nitrate; nitrite; neuromuscular; taekwondo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice supplementation (Experimental): 140 mL of beetroot juice (12.8 mmol of NO3-, Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) made from concentrates of beetroot juice (98%) and lemon juice (2%) (nutritional information (per 100 mL), energy: 373 kJ; fat: 0 g; carbohydrates: 18 g [sugars: 17 g]; protein: 3.7 g; salt: 0.48 g)
  Interventions: Dietary Supplement: Beetroot juice (James White, UK)
- Placebo supplementation (Placebo Comparator): 140 mL of beetroot juice placebo without nitrates (0.08 mmol of NO3-, Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) made from concentrates of beetroot juice (98%) and lemon juice (2%) (nutritional information (per 100 mL), energy: 373 kJ; fat: 0 g; carbohydrates: 18 g [sugars: 17 g]; protein: 3.7 g; salt: 0.48 g)
  Interventions: Dietary Supplement: Placebo acute supplementation (James White, UK)

INTERVENTIONS:
Dietary Supplement: Beetroot juice (James White, UK) — One serving 140 mL of BJ (12.8 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) after an overnight fast and 2.5 h before initiating the testing session.
  Arms: Beetroot juice supplementation
Dietary Supplement: Placebo acute supplementation (James White, UK) — One serving 140 mL of BJ (0.04 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) after an overnight fast and 2.5 h before initiating the testing session.
  Other Names: Beetroot juice placebo
  Arms: Placebo supplementation

SUMMARY:
Beetroot juice is a good source of nitrate (NO3-), which is a precursor of nitric oxide (NO) through the NO3- to nitrite (NO2-) to NO pathway (Lundberg et al., 2008). Consequently, it is thought that a minimum threshold may exist for dietary NO3- consumption of at least 5 mmol to enhance athletic performance (Senefeld et al., 2020). In turn, systematic reviews have documented that the use of beetroot juice supplementation enhances muscle strength and power-related attributes (Gonzalez et al., 2023), as well as performance in repeated high-intensity activity bouts (Alsharif et al., 2023; Dominguez et al., 2018). However, beetroot juice supplementation has been shown to have equivocal effects on neuromuscular performance specifically among individual sport athletes (e.g. taekwondo). Thus, the aim of this study was to determine the effects of acute beetroot juice ingestion (140 mL, 12.8 mmol NO3-) on neuromuscular performance in elite female taekwondo athletes.

DETAILED DESCRIPTION:
Beetroot juice is a good source of nitrate (NO3-), which is a precursor of nitric oxide (NO) through the NO3- to nitrite (NO2-) to NO pathway (Lundberg et al., 2008). This pathway is thought to promote increased sarcoplasmic reticulum calcium release and re-uptake with ensuing enhancements in force output within type II muscle fibers (Hernandez et al., 2012), as well as increased neurotransmitter release (Esen et al., 2022) and attenuated muscle potassium efflux (Wylie et al., 2013) that could benefit neuromuscular performance. Consequently, it is thought that a minimum threshold may exist for dietary NO3- consumption of at least 5 mmol to enhance athletic performance (Senefeld et al., 2020). In turn, systematic reviews have documented that the use of beetroot juice supplementation enhances muscle strength and power-related attributes (Gonzalez et al., 2023), as well as performance in repeated high-intensity activity bouts (Alsharif et al., 2023; Dominguez et al., 2018). However, beetroot juice supplementation has been shown to have equivocal effects on neuromuscular performance specifically among individual sport athletes (e.g. taekwondo). Thus, the aim of this study was to determine the effects of acute beetroot juice ingestion (140 mL, 12.8 mmol NO3-) on neuromuscular performance in elite female taekwondo athletes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 to 40 years
* Competed in international taekwondo competitions representing her national teams.
* More than6 years of training experience (at least 3 sessions per week).
* Female taekwondo athletes.

Exclusion Criteria:

* Male taekwondo athletes.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Simulated taekwondo Combat (actions/time) | 1-week
  Simulated taekwondo combat were performed according to the guidelines of the World Taekwondo (WT), and participants were divided based in the Olympic weight categories (WT, 2016). All the combats were executed in an official octagonal and homologated competition area while an international referee (who doesn´t know the experimental treatments) arbitrated. Today the rules of WTF led to use electronic protectors as protecting of athletes and identify electronically the punctuations (Del Vecchio, Franchini, Del Vecchio, & Pieter, 2011). Variables analyzed were attack time (AT), step time (ST), pause time (PT), period without attack (PWA = ST+PT), numbers of attacks (AN), the ratio for attack time and step time (R1 = AT/ST), and ratio for action time and step time (R2 = (AT+ST) /PT).

SECONDARY OUTCOMES:
Changes in maximal jump height (cm) | 1-week
  Maximal jump height using a contact platform
Reaction time (ms) | 1-week
  Reaction times in a specific reaction test with BlazePod ((Play Coyotta Ltd., Tel Aviv, Israel)
Blood lactate concentrations (mmol·L-1) | 1-week
  Previous to the warm-up, just to the end of the simulated combat, and 3 minutes after, a researcher extracted a blood sample of the pad of the index finger of the left hand of the participants.
Rating of percevied exertion (RPE) (measured using scale 6-20 points) | 1-week
  Immediately after each one of the 3 assaults, participants were asked for providing her RPE using a Borg scale from 6 to 20 points

CONTACTS AND LOCATIONS:
Locations (1):
- Universida Pontificia Comillas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No